CLINICAL TRIAL: NCT02276625
Title: One-visit Multi-site Pre-exposure Intradermal Rabies Vaccination: Dose Finding in Healthy Adults.
Brief Title: One-visit Multi-site Intradermal Rabies Vaccination - Dose Finding
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R5
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Rabies Pre-exposure Prophylaxis
MeSH Terms: interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A - ID (Experimental): Intradermal administration. 20% dose in a single visit.
  Interventions: Biological: rabies vaccine
- B - ID (Experimental): Intradermal administration. 40% dose in a single visit.
  Interventions: Biological: rabies vaccine
- C - ID (Experimental): Intradermal administration. 60% dose in a single visit.
  Interventions: Biological: rabies vaccine
- D - IM (Active Comparator): 1x IM
  Interventions: Biological: rabies vaccine

INTERVENTIONS:
Biological: rabies vaccine — Compare ID administration to IM administration. 1 visit schedule.

SUMMARY:
To determine optimum dose level for a single visit multidose intradermal injection of rabies vaccine with the aim to induce immunological memory in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Good health according to the investigator
* Willingness and ability to adhere to the study regimen
* Able to give informed consent

Exclusion Criteria:

* Known or suspected previous vaccination against rabies
* Known or suspected allergy against any of the vaccine components
* History of unusual or severe reactions to any previous vaccination
* Immunocompromized state due to illness or medication
* Administration of plasma or blood products three months prior to inclusion in the study
* (hydroxy)chloroquine or mefloquine use
* History of any neurological disorder including epilepsy or febrile seizures
* Pregnancy or breastfeeding
* Any current infectious disease other than seasonal cold
* Bleeding disorders or use of anticoagulants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Memory response in vaccinated subjects 1 year after primary vaccination (defined as seroprotection rate for all subjects within 7 days post-booster in a simulated post-exposure scenario) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Leo Visser, M, PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands